CLINICAL TRIAL: NCT02529956
Title: A Randomized, Subject-blind, Investigator-blind, Placebo-controlled, Single-dose, Dose-escalating Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of UCB4940 in Patients With Mild to Moderate Psoriasis
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of UCB4940 in Patients With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP0008; 2012-002086-35 (EudraCT Number)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Mild to Moderate Psoriasis
Keywords: Psoriasis; UCB4940
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- UCB4940 8 mg (Experimental): Single intravenous (iv) infusion of UCB4940 8 mg over at least 60 minutes.
  Interventions: Drug: UCB4940
- UCB4940 40 mg (Experimental): Single intravenous (iv) infusion of UCB4940 40 mg over at least 60 minutes.
  Interventions: Drug: UCB4940
- UCB4940 160 mg (Experimental): Single intravenous (iv) infusion of UCB4940 160 mg over at least 60 minutes.
  Interventions: Drug: UCB4940
- UCB4940 480 mg (Experimental): Single intravenous (iv) infusion of UCB4940 480 mg over at least 60 minutes.
  Interventions: Drug: UCB4940
- UCB4940 640 mg (Experimental): Single intravenous (iv) infusion of UCB4940 640 mg over at least 60 minutes.
  Interventions: Drug: UCB4940
- Placebo (Placebo Comparator): Single intravenous (iv) infusion of Placebo over at least 60 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UCB4940 — * Active Substance: UCB4940
  * Pharmaceutical Form: Solution for infusion
  * Concentration: 80 mg/ml
  * Route of Administration: Intravenous use
  Arms: UCB4940 160 mg; UCB4940 40 mg; UCB4940 480 mg; UCB4940 640 mg; UCB4940 8 mg
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Solution for infusion
  * Concentration: 0.9 % sodium chloride aqueous solution
  * Route of Administration: Intravenous use
  Arms: Placebo

SUMMARY:
To evaluate the safety of UCB4940 administered by iv infusion of a single ascending dose in subjects with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Subject is male or female, aged ≥ 18 years to ≤ 70 years at Screening. Female subjects must either be postmenopausal (at least 1 year), permanently sterilized or, if of childbearing potential, must be willing to use at least 2 effective methods of contraception, including a barrier method during the study period. Effective methods of contraception are methods of birth control, which result in a low failure rate when used consistently and correctly, such as implants, injectables, oral contraceptives, progesterone-releasing intrauterine systems or the TCu 380A intrauterine device, complete sexual abstinence, or vasectomized partner. Male subjects with partners of childbearing potential must be willing to use a condom when sexually active. Both male and female subjects must use the above mentioned contraception for 20 weeks after administration of study drug (anticipated 5 half-lives)
* Subject has had a confirmed diagnosis of mild to moderate plaque-type psoriasis for at least 6 months involving ≤ 5 % of body surface area (BSA) (excluding the scalp)
* Subject has a body mass index of ≤ 35 kg/m^2 at Screening
* Subject has a minimum of 2 psoriatic lesions with at least 1 plaque in a site suitable for biopsy

Exclusion Criteria:

* Female subject who is pregnant, or plans to become pregnant during the study, or lactating, or sexually active with childbearing potential who is not using a medically accepted birth control method
* Subject has received systemic nonbiologic psoriasis therapy (methotrexate [MTX], steroids, cyclophosphamide) or psoralen plus ultraviolet A (PUVA)/ultraviolet A (UVA) phototherapy within 4 weeks prior to Screening
* Subject has received treatment with biologic agents within 12 months prior to the study
* Subject has received live attenuated vaccination within 6 weeks prior to Screening or intends to have such a vaccination during the course of the study
* Subject has received any investigational drug or experimental procedure within 90 days or 5 half-lives, whichever is longer, prior to IMP administration
* Subject requires treatment with a nonsteroidal anti-inflammatory drug during the study period. Paracetamol will be permitted for use as an antipyretic and/or analgesic
* Subject has an active infection (eg, sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to IMP administration. When in doubt, the Investigator should confer with the UCB Study Physician
* Subject has a history of a positive tuberculosis (TB) test or evidence of possible TB or latent TB infection at Screening that cannot be attributed to a prior Bacillus Calmette-Guérin inoculation
* Subject has renal or liver impairment, defined as:

  * For women, serum creatinine level ≥ 125 μmol/L; for men, ≥ 135 μmol/L, or
  * ALT and aspartate aminotransferase ≥ 2x ULN, or
  * Alkaline phosphatase and bilirubin > 1.5x ULN (an isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35 %)
* Subject has active neoplastic disease or history of neoplastic disease within 5 years of Screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting at least 1 Treatment-Emergent Adverse Event (TEAE) during the Treatment Period (20 Weeks) | Baseline to 20 Weeks
Number of subjects prematurely discontinuing due to a Treatment-Emergent Adverse Event (TEAE) during the Treatment Period (20 Weeks) | Baseline to 20 Weeks
Number of subjects reporting at least 1 Serious Adverse Event (SAE) during the Treatment Period (20 Weeks) | Baseline to 20 Weeks

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Area under the plasma concentration-time curve from time 0 to infinity (AUC(0-inf)) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Area under the plasma concentration-time curve from time 0 to the time of last quantifiable concentration (AUC(0-t)) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Time to reach Cmax (Tmax) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Terminal elimination half-life (t1/2) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
First order terminal elimination rate constant (λz) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Total body clearance (CL) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Volume of distribution in terminal phase (Vz) | Pharmacokinetic samples will be taken predose and 0-48 hr post-dose, 72 hr post-dose, 96 hr post-dose, Week-1 through Week-20
Percentage Change from Baseline to Week 12 in the Lesion Severity Score (LSS) | Baseline to Week 12
Percentage Change from Baseline to Week 12 in thickness of the plaque | Baseline to Week 12
Percentage Change from Baseline to Week 12 in lesion area | Baseline to Week 12
Percentage Change from Baseline to Week 12 in Psoriasis Area and Severity Index (PASI) | Baseline to Week 12
Percentage Change from Baseline to Week 12 in Physician's Global Assessment (PGA) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 8229493 (UCB)
Locations (1):
- 1, Harrow, United Kingdom

REFERENCES:
- [Derived] Glatt S, Helmer E, Haier B, Strimenopoulou F, Price G, Vajjah P, Harari OA, Lambert J, Shaw S. First-in-human randomized study of bimekizumab, a humanized monoclonal antibody and selective dual inhibitor of IL-17A and IL-17F, in mild psoriasis. Br J Clin Pharmacol. 2017 May;83(5):991-1001. doi: 10.1111/bcp.13185. Epub 2017 Jan 10. PMID 27859546